CLINICAL TRIAL: NCT00630760
Title: A Multiple-Center, Open-Label, Dose Escalation Study of the Safety and Pharmacokinetics of Oral NRX 194204 Capsule Administered Daily for a Minimum of 4 Weeks in Patients With Refractory Malignancies
Brief Title: Oral NRX 194204 in Patients With Refractory Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew study. Accrual not completed
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-07-6
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Refractory Malignancies
MeSH Terms: conditions — Neoplasms | interventions — AGN 194204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): NRX 194204 capsules in escalating doses, starting at 3mg/m2.
  Interventions: Drug: NRX 194204

INTERVENTIONS:
Drug: NRX 194204 — NRX 194204 capsules given 3mg/m2 daily x 28 days. Repeated until PD

SUMMARY:
This phase I study will determine the safety profile of NRX 194204 on this schedule; it will evaluate the pharmacokinetic profile of NRX 194204 in cancer patients; and will investigate anti-tumor activity as manifested by standard response criteria, or by tumor markers.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Histologically confirmed cancer refractory to conventional therapy or refractory cancer for which there is no known effective or standard therapy.
* Measurable or non-measurable disease.
* Male or female, 18 to 75 years of age, inclusive.
* ECOG Performance Status 0-2
* Life expectancy greater than 24 weeks.
* Able to swallow the oral capsule form of the drug.
* Hematology: Hemoglobin greater than or equal to 8.5; Platelets greater than or equal to100,000; Neutrophils greater than or equal to 1500
* PT and PTT within normal limits, except for patients receiving oral Vitamin K antagonist for thromboembolic prophylaxis, in whom an INR less than 2 is allowable.
* Biochemistry: Total bilirubin less than or equal to 1.5 x ULN; AST/ALT less than or equal to 3.0 x ULN; Serum creatinine less than or equal to 2.0 mg/dl; Serum calcium less than or equal 11.5 mg/dl; Fasting serum triglycerides less than or equal 2.5 x ULN
* Endocrine: Thyroid stimulating hormone (TSH)within institutional normal limits (typically greater than 0.5 mU/L and less than 5.5 mU/L)
* Negative urine pregnancy test for women of child-bearing potential at screening and on Day 0, and agreement to use two reliable forms of contraception during therapy and for 1 month following discontinuation of therapy unless abstinence is the chosen birth control method.
* Able to follow study instructions, accessible for treatment and follow-up, and likely to complete all study requirements

Exclusion Criteria:

* Major surgery within previous 4 weeks; large field radiation therapy or chemotherapy ,including investigational agents or participation in another clinical study within previous 3 weeks; mitomycin C or nitrosoureas within 6 weeks. In all instances patients must have fully recovered from acute toxicities related to prior therapies.
* Systemic retinoid therapy, or large doses of Vitamin A during previous 4 weeks.
* Patients with any prior or current history of thyroid disease, with any history of pituitary disease, or with any history of prior or current treatment with thyroid replacement hormone.
* Primary brain tumors, active brain metastasis including progression from last scan or evidence of cerebral edema, or clinical symptoms of brain metastasis. Patients with prior history of brain metastasis must have brain imaging performed and be found to be stable or improving over a minimum interval of 8 weeks.
* Requirement for steroids. Note:Patients taking stable dosages of GnRH analogues or Megace for at least the previous 3 months will be allowed into the study.
* Current enrollment in an investigational drug or device study or participation in such a study within 21 days of entry into this study.
* Prior enrollment in the study (Quest 194204-101-00); patients may only enroll once and be treated only at one dose level.
* Known sensitivity to any of the ingredients in the study medication.
* Known HIV-positive patients.
* Females who are pregnant, nursing, or planning a pregnancy.
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with absorption of study medication.
* Clinically significant abnormalities on screening ECG (QTc greater than 480 msec).
* Patient has a condition or is in a situation that, in the investigator's opinion, may put him/her at significant risk, may confound the study results, or may interfere significantly with his/her participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine MTD | Weekly

SECONDARY OUTCOMES:
Efficacy | Day 29 and then every 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States